CLINICAL TRIAL: NCT04440111
Title: Teaching Children Basic Life Support: Randomized Clinical Trial
Brief Title: Basic Life Support by Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cristina Genzor (Other)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Sponsor-Investigator, Cristina Genzor, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PI19/490
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Cardiopulmonary Arrest With Successful Resuscitation; Child, Only

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): One year basic life support training
  Interventions: Other: One year training
- Experimental group (Sham Comparator): Two years basic life support training
  Interventions: Other: Two years training

INTERVENTIONS:
Other: One year training — At first, children will make a test to evaluate their pre- intervention basic support life knowledge.
  Secondly, they will receive a theoretical class about BLS, based on European Resuscitation Council Guide 2015.
  After that, they will make a practical workshop on BLS. Finally they will repeat the initial test. The second year, this group will only make the test, they won't receive any theory or practice.
  Other Names: One year basic life support training
  Arms: Control group
Other: Two years training — At first, children will make a test to evaluate their pre- intervention basic support life knowledge.
  Secondly, they will receive a theoretical class about BLS, based on European Resuscitation Council Guide 2015. After that they will make a practical workshop on BLS.
  Finally they will repeat the initial test. The second year, this group will repeat the same process.
  Other Names: Two years basic life support training
  Arms: Experimental group

SUMMARY:
A controlled clinical trial will be performed.

School children from the age of 10 to 11 will be selected to learn basic life support (BLS) in a primary school of Zaragoza.

One of the groups will learn BLS in two consecutive years and the other group will learn BLS only the first year.

The investigators think that the knowledge will be better in the group that receives two interventions.

DETAILED DESCRIPTION:
A controlled clinical trial will be performed.

72 participants between 10 and 11 years old will be selected and randomized to participate.

Control group and experimental group will enrolled 36 participants each one. Control group will receive BLS training once. Experimental group will receive BLS training in two consecutive years.

Previous and after training a test will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Children from 10 to 12 years old that are attending to the selected school at the moment of the intervention
* Children with signed consent given by parents at the moment of the intervention

Exclusion Criteria:

* Children not attending all the theorical and practical interventions
* Children not completing all test.
* Children with learning disabilities

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the knowledge level of BLS after receiving one or two interventions | 3 hours
  A questionnaire will be performed. It will consist of a 14 multiple-choice questions. Each question will have 4 choices, one of wich will be correct. Questions will be based on the European Resuscitation Council (ERC) Guidelines 2015.
To compare test results obtained previous and after intervention. | 1 month
  A questionnaire will be performed. It will consist of a 14 multiple-choice questions. Each question will have 4 choices, one of wich will be correct. Questions will be based on the European Resuscitation Council (ERC) Guidelines 2015. After obteining the marks, the results will be compared using Statistical Analysis Software.

CONTACTS AND LOCATIONS:
Locations (1):
- Cristina Genzor Ríos, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Semeraro F, Wingen S, Schroeder DC, Ecker H, Scapigliati A, Ristagno G, Cimpoesu D, Bottiger BW. KIDS SAVE LIVES-Three years of implementation in Europe. Resuscitation. 2018 Oct;131:e9-e11. doi: 10.1016/j.resuscitation.2018.08.008. Epub 2018 Aug 8. No abstract available. PMID 30098386
- [Result] Bottiger BW, Van Aken H. Kids save lives--Training school children in cardiopulmonary resuscitation worldwide is now endorsed by the World Health Organization (WHO). Resuscitation. 2015 Sep;94:A5-7. doi: 10.1016/j.resuscitation.2015.07.005. Epub 2015 Jul 21. No abstract available. PMID 26209417
- [Result] Bohn A, Van Aken HK, Mollhoff T, Wienzek H, Kimmeyer P, Wild E, Dopker S, Lukas RP, Weber TP. Teaching resuscitation in schools: annual tuition by trained teachers is effective starting at age 10. A four-year prospective cohort study. Resuscitation. 2012 May;83(5):619-25. doi: 10.1016/j.resuscitation.2012.01.020. Epub 2012 Jan 28. PMID 22286049
- [Result] Lukas RP, Van Aken H, Molhoff T, Weber T, Rammert M, Wild E, Bohn A. Kids save lives: a six-year longitudinal study of schoolchildren learning cardiopulmonary resuscitation: Who should do the teaching and will the effects last? Resuscitation. 2016 Apr;101:35-40. doi: 10.1016/j.resuscitation.2016.01.028. Epub 2016 Feb 8. PMID 26868079
- [Result] Bohn A, Lukas RP, Breckwoldt J, Bottiger BW, Van Aken H. 'Kids save lives': why schoolchildren should train in cardiopulmonary resuscitation. Curr Opin Crit Care. 2015 Jun;21(3):220-5. doi: 10.1097/MCC.0000000000000204. PMID 25922895
- [Result] Haseneder R, Skrzypczak M, Haller B, Beckers SK, Holch J, Wank C, Kochs E, Schulz CM. Impact of instructor professional background and interim retesting on knowledge and self-confidence of schoolchildren after basic life support training: a cluster randomised longitudinal study. Emerg Med J. 2019 Apr;36(4):239-244. doi: 10.1136/emermed-2018-207923. Epub 2019 Feb 16. PMID 30772830